CLINICAL TRIAL: NCT00345384
Title: Post-Operative Infusion of Low-Dose Dexmedetomidine for the Control of Post-Operative Pain in Thoracotomy Patients: A Randomized, Double-Blind, Controlled Pilot Study
Brief Title: Dexmedetomidine for the Control of Post-Operative Pain in Thoracotomy Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 005-201
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Post-operative Pain; Respiratory Depression
Keywords: Dexmedetomidine; Sedation; Opioid; Respiratory depression
MeSH Terms: conditions — Pain, Postoperative; Respiratory Insufficiency | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): One group (placebo comparator) will receive a normal saline infusion, set at a rate as if it were the active drug.
  Interventions: Other: Placebo (Normal Saline)
- Dexmedetomidine (Active Comparator): The second group (the study group) will receive a continuous infusion of dexmedetomidine titrated from 0.1 - 0.5 mics/kg/h to control pain for up to 24 hours after they are admitted to an open nursing unit after discharge from the PACU or ICU
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine titrated over 24 hours
  Other Names: Precedex, Dexdor Titrated 0.1 to 0.5 ug.kg.h-1
  Arms: Dexmedetomidine
Other: Placebo (Normal Saline)
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, hemodynamic and respiratory stability of a low-dose of dexmedetomidine infusion in post-operative surgical in-patients undergoing thoracic surgery after discharge from PACU or ICU.

DETAILED DESCRIPTION:
Dexmedetomidine has sedative and analgesic properties that may reduce the opioid requirement in post-operative patients, thereby decreasing the chance of post-operative respiratory depression that occurs with opioid administration. In addition, patients may be more alert with less opioid medication. Currently, dexmedetomidine is not approved for use longer than twenty-four hours and must only be administered in the Intensive Care Unit where patients can be continuously monitored.

This is a prospective, double-blinded, control group pilot study. One group (the control group) will receive a normal saline infusion and the second group (the treatment group) will receive low-dose Dexmedetomidine for up to 24 hours after they are admitted to an open nursing unit (not an Intensive Care Unit).

During the surgery, the anesthesiologist will administer dexmedetomidine during the surgical procedure after an optional loading dose. All patients will receive pain medication using a Patient Controlled Analgesia (PCA) pump as per standard practice. In addition, if the physician deems necessary, an On-Q Pain Pump will deliver local anesthetic surrounding the incision under direction of the surgeon.

Before discharge from the PACU or ICU, each subject will receive either low-dose dexmedetomidine or normal saline using a continuous infusion pump for up to 24 hours after the subject is discharged from either the PACU or the ICU to an open nursing unit. While on the open nursing unit patient vital signs, oxygen saturation, Ramsay score and pain score will recorded every two hours until the treatment drug is stopped.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I, II or III
* Undergoing thoracic surgery on an inpatient basis
* Age 18 up to 85 years of age

Exclusion Criteria:

* Subject is pregnant and/or lactating
* Subject has a serious Central Nervous System (CNS)pathology/trauma that, per clinical judgment of the investigator, precludes responsiveness or survival.
* Subject for whom alpha-2 agonists are contraindicated
* Subject meets any of the following cardiovascular criteria:
* Acute unstable angina (defined during current hospital stay)
* Suspicion of acute myocardial infarction.
* Considered to have a left ventricular ejection fraction of less than 30%.Decision to exclude is predicated in the Investigator's opinion, and may be based on any combination of acute presentations, recently preformed diagnostic studies, or a history that suggests poor cardiac function. Pulmonary congestion of a non-cardiac origin or mild congestive failure primarily attributable to etiologies other than poor ventricular function are not exclusion criteria.
* Subject has participated in a trial with any experimental drug within 30 days prior to enrollment in the study, or has ever been enrolled in this study.
* Subject is unable to undergo any procedures required by the protocol.
* Subject has acute hepatitis, a history or presence of chronic hepatitis, and /or has had a positive result for Hepatitis B surface antigen test.
* Subject requires dialysis (e.g., hemodialysis, peritoneal dialysis, CVVHD).
* Subject has a known, uncontrolled seizure disorder.
* Subject has a known psychiatric illness that could confound a normal response to sedative treatment.
* Subject is terminally ill with a life duration expectancy of < 60 days.
* Subject has a history of Obstructive Sleep Apnea.
* Oxygen saturation is < 90% on room air.
* Subject is on beta blocker medication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramsay, MD, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center - Department of Anesthesiology, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited from the from the BUMC Operating Room schedule prior to their procedure. Informed consent will be obtained in a secure area. Recruitment will continue until goal reached.
Pre-assignment Details: Participants were required to be between the ages of 18-85 and receiving general anesthesia with an AMerican Society of Anesthesiologists score of three or less, and undergoing thoracotomy surgery. Liver and renal failure patients were excluded.
Groups:
- Normal Saline: Blinded Normal saline infusion titrated as if study drug
- Dexmedetomidine: Received Dexmedetomidine for 24 hours
Period: Overall Study
Arm/Group | Normal Saline | Dexmedetomidine
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 13 were withdrawn from study prior to initiation of drug due to exclusion criteria that required an overnight stay in Recovery or ICU.
Groups:
- Normal Saline: Standard of care
- Dexmedetomidine: titrated IV for 24 hours post ICU
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Dexmedetomidine | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.8) | 61 (10.75) | 60 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Measure Any Reduction in the Amount of Opioid Administered to Patients in the Dexmedetomidine Study Arm.
Description: To measure the amount of opioid use requested by patients enrolled in the dexmedetomidine study arm during the observation period of 24 hours, up to 30 hours per patient.
Time Frame: An average of 24 hours, up to 30 hours per patient
Population: Participants completing the study were analyzed as per protocol
Measure: Number (95% Confidence Interval); unit: IV morphine equivalency in mg
Groups:
- Placebo: Patient group to receive placebo (saline).
- Dexmedetomidine: Patient group to receive Dexmedetomidine.
Arm/Group | Placebo | Dexmedetomidine
Number analyzed (Participants) | 19 | 19
IV morphine equivalency in mg
  Morphine equivalency administered | 49 [14 to 84] | 29 [3 to 55]
  Adjusted for total time on study drug | 54 [17 to 91] | 35 [7 to 63]
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine; Test type: Superiority or Other; p = 0.03, t-test, 2 sided; Precentage Difference = 41 — The percentage in opioid use by the dexmedetomidine group in comparison to the placebo for the period of time on study drug is calculated as follows: numerator = 29, denominator = 49
Statistical Analysis 2: Comparison: Placebo vs Dexmedetomidine; Test type: Superiority or Other; p = 0.04, t-test, 2 sided; Percentage difference = 35 — A measure of opioid use, weighted for total time on study drug. This is examined by a comparison of the dexmedetomidine group to the placebo group: numerator = 35, denominator = 54

2. Secondary Outcome: Measure the Amount of Respiratory Depression in Each Groups
Description: Respiratory depression and deep levels of sedation can occur when morphine patient-controlled analgesia is prescribed for postoperative patients. In this secondary outcome measure, it was hypothesized that the addition of a dexmedetomidine infusion to the postoperative pain management protocol would reduce the amount of morphine delivered by a PCA pump while providing adequate analgesia. Data are reported for the time period 6 to 16 hours. However, the subjects were on the study for an average of 24 hours, up to 30 hours.
Time Frame: Hours 6 to 16
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo: Control group to receive a normal saline infusion, set at a rate as if it were the active drug.
- Dexmedetomidine: Study group to receive a continuous infusion of dexmedetomidine titrated from 0.1 - 0.5 mics/kg/h to control pain for up to 30 hours after they are admitted to an open nursing unit after discharge from the PACU or ICU
  Dexmedetomidine: Dexmedetomidine titrated over 24 hours
Arm/Group | Placebo | Dexmedetomidine
Number analyzed (Participants) | 19 | 19
mmHg | 45 (9) | 42 (8)
Statistical Analysis 1: Comparison: Placebo vs Dexmedetomidine; The p-value reported in this table corresponds with the 6 to 16 hour time frame; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 week from initiation of study drug.
Description: 0 serious adverse events were detected in patients enrolled in this study.
Groups:
- Normal Saline Group: Normal saline infused at calculated rate as if it were study drug
- Study Drug Group: Dexmedetomidine titrated IV from 0.1 microgram/kg/h upto 0.5 microgram/kg/h to control pain for 24 hours post ICU
Arm/Group | Normal Saline Group | Study Drug Group
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline Group (N=19) | Study Drug Group (N=19)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) — systolic BP < 90 Mm Hg
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) — heart rate < 50 bpm
Tacycardia (Cardiac disorders) | 3 (3) | 1 (1) — Heart rate > 110 bpm

LIMITATIONS AND CAVEATS:
Pilot study with small numbers of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No